CLINICAL TRIAL: NCT05312736
Title: Gyrate Atrophy Ocular and Systemic Study
Acronym: GYROS
Status: Active, not recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Conquering Gyrate Atrophy Foundation (Unknown); Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: GYROS; R01FD007628 (FDA)
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-08

CONDITIONS: Gyrate Atrophy; Gyrata of Choroid and Retina; Atrophy; Ornithine-δ-aminotransferase; OAT; Chorioretinal Degeneration
Keywords: Gyrate Atrophy; OAT
MeSH Terms: conditions — Gyrate Atrophy; Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vision Cohort 1: Criteria that must be met in the better eye* at the Screening Visit:
  visual acuity ETDRS letter score of 54 or more (approximate Snellen equivalent 20/80 or better) and visual field** diameter 10 degrees or more in every meridian of the central field
  The better eye is defined as the eye with the better Screening Visit ETDRS visual acuity. However, if both eyes have the same visual acuity, which is defined as the same Snellen equivalent, then the determination will be made at investigator discretion. In this scenario, the investigator will consider the eye with better fixation or clearer ocular media to permit highest quality retinal imaging.
  The visual field (VF) is defined as the clinically determined kinetic VF III4e performed within the last 18 months prior to the Screening Visit or performed on the day of the Screening Visit.
- Vision Cohort 2: Criteria that must be met in the better eye* at the Screening Visit:
  visual acuity ETDRS letter score of 19-53 (approximate Snellen equivalent 20/100 - 20/400) OR visual acuity ETDRS letter score of 54 or more (approximate Snellen equivalent 20/80 or better) and visual field** diameter less than 10 degrees in any meridian of the central field.
  The better eye is defined as the eye with the better Screening Visit ETDRS visual acuity. However, if both eyes have the same visual acuity, which is defined as the same Snellen equivalent, then the determination will be made at investigator discretion. In this scenario, the investigator will consider the eye with better fixation or clearer ocular media to permit highest quality retinal imaging.
  The visual field (VF) is defined as the clinically determined kinetic VF III4e performed within the last 18 months prior to the Screening Visit or performed on the day of the Screening Visit.
- Vision Cohort 3: Criteria that must be met in the better eye* at the Screening Visit:
  visual acuity ETDRS letter score of 18 or less (approximate Snellen equivalent 20/500 or worse).
  The better eye is defined as the eye with the better Screening Visit ETDRS visual acuity. However, if both eyes have the same visual acuity, which is defined as the same Snellen equivalent, then the determination will be made at investigator discretion. In this scenario, the investigator will consider the eye with better fixation or clearer ocular media to permit highest quality retinal imaging.
  The visual field (VF) is defined as the clinically determined kinetic VF III4e performed within the last 18 months prior to the Screening Visit or performed on the day of the Screening Visit.

SUMMARY:
The Gyrate Atrophy Ocular and Systemic Study characterizes the natural history of ornithine levels and retinal degeneration (RD) associated with disease-causing OAT variants in the presence of standard care dietary treatment regimens over 4 years. The research goal is to understand the impact of OAT mutations on plasma ornithine levels and retinal degeneration. Funding Source- FDA OOPD

DETAILED DESCRIPTION:
Gyrate atrophy is a rare inherited chorioretinal degeneration that is associated with hyperornithinemia, an inborn error of metabolism caused by autosomal recessive mutations in the ornithine aminotransferase (OAT) gene. Gyrate atrophy is characterized by childhood-onset nyctalopia and sharply demarcated areas of chorioretinal atrophy that initially involve the midperipheral fundus. The atrophic areas typically coalesce and enlarge towards the posterior pole in the second and third decades of life, leading to severe visual field constriction and vision loss if left untreated. The current standard care treatment of gyrate atrophy is an arginine restricted diet that is implemented in practice using dietary protein restriction with essential amino acid supplementation. However, dietary treatment is highly burdensome on patients and negatively impacts quality of life such that only about ~20% of patients are able to comply. Strict adherence to dietary protein restriction (particularly through adolescence), essential amino acid supplementation, and nutritional management of body weight especially during intercurrent illness and pregnancy are among the challenges of treatment. Periods of suboptimal dietary control led to plasma ornithine elevation and progressive chorioretinal degeneration.

Investigators are developing gene therapy as a potential one-time treatment that could arrest disease progression while avoiding or reducing the need for dietary treatment. To facilitate a future interventional gene therapy clinical trial, there is a need to evaluate natural history of and the relationship between potential clinical trial outcome measures.

The objectives of the OAT gene natural history study are as follows:

1. Natural History

   1. Characterize the natural history of retinal degeneration associated with disease-causing OAT variants in the presence of standard care dietary treatment regimens over four (4) years, using functional, structural, and patient-reported outcome measures.
   2. Characterize the natural history of ornithine levels associated with disease-causing OAT variants in the presence of standard care dietary treatment regimens over four (4) years.
   3. Determine within-patient variability of ornithine levels associated with disease-causing OAT variants in the presence of standard care dietary treatment regimens over four (4) years.
   4. Evaluate inter-eye correlation on ocular measures.
2. Metabolic-Structure-Function Relationships

   1. Explore relationship of structural outcomes with functional outcomes in individuals with disease-causing OAT variants.
   2. Explore relationship of plasma ornithine levels with structural and functional outcomes in individuals with disease-causing OAT variants.
3. Identify Rapid Progressors

   1. Explore possible risk factors (genotype, phenotype, environmental, comorbidities, and dietary therapy/supplements) for progression of the functional, structural, and patient-reported outcome measures over four (4) years in individuals with disease-causing OAT variants.
   2. Explore possible risk factors (genotype, phenotype, environmental, comorbidities, and dietary therapy/supplements) for ornithine levels over four (4) years in individuals with disease-causing OAT variants.

The expected impact of the OAT gene natural history study is to inform a future interventional clinical trial design and implementation, including the following:

1. Determine within-patient variability of ornithine levels.
2. Develop quantitative measures of progression of the area of preserved retina and establish its reproducibility, sensitivity to change, and relationship with other measures.
3. Establish rates of progression of retinal degeneration on all functional, structural, and patient-reported outcome measures, and determine which measures are most sensitive to change.
4. Determine primary time points and duration for a planned future treatment trial.
5. Use variability and inter-eye correlation of outcomes for trial sample size calculations.
6. Identify candidates for the future trial, including eligibility criteria based on risk factors and cut points for severity of disease most likely to benefit from treatment.
7. Establish study procedures and workflows for practical implementation of the same testing procedures in a future trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all the following inclusion criteria at the Screening Visit in order to be eligible to enroll into the genetic screening phase.
* Willing to participate in the study and able to communicate consent during the consent process.
* Willing and able to complete all study visit assessments at each visit over the forty-eight (48) month study period. Age ≥ 12 years.

Must meet one (1) of the Genetic Screening Criteria below:

* At least 2 disease-causing variants in the OAT gene which are homozygous or heterozygous in trans, based on a report from a clinically certified lab, or a report from a research lab that has been pre-approved by the study Genetics Committee.
* At least 2 disease-causing variants in the OAT gene with unknown phase, based on a report from a clinically certified lab, or a report from a research lab that has been pre-approved by the study Genetics Committee, AND must meet both of the following phenotype criteria: .Classic fundus appearance of gyrate atrophy (based on investigator discretion) AND Elevated ornithine levels >300 μmol/L (documented on any prior lab report).

Note: if a participant has a variant(s) of unknown significance, they will still qualify if they meet the Genetic Screening Criteria above. Ocular Inclusion Criteria Participant must meet the following criteria at the Screening Visit to enroll into the genetic screening phase.

Both eyes must have a clinical diagnosis of retinal dystrophy. Both eyes must permit good quality photographic imaging (e.g., but not limited to, clear ocular media, adequate pupil dilation, stable fixation).

Exclusion Criteria:

* Participants must not meet any of the following exclusion criteria at the Screening Visit in order to be eligible to enroll into the genetic screening phase.
* Single pathogenic or likely pathogenic genetic variants known to be associated with autosomal dominant retinitis pigmentosa/retinal dystrophy (AD, heterozygous), X-374 linked retinitis pigmentosa/retinal dystrophy (XL, hemizygous), or mitochondrial inheritance.
* Expected to enter experimental treatment trial at any time during this study. History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy, including hydroxychloroquine, chloroquine, thioridazine, and deferoxamine. Note: Since this is a Natural History Study collecting data on the progression of Gyrate Atrophy, pregnant women will not be specifically excluded from participation.

Ocular Exclusion Criteria:

* If either eye has any of the following ocular exclusion criteria at the Screening Visit, then the participant is not eligible to enroll into the genetic screening phase.
* Current vitreous hemorrhage.
* Current or any history of tractional or rhegmatogenous retinal detachment.
* Current or any history of (for example, but not limited to prior to cataract or refractive surgery) spherical equivalent of the refractive error worse than -8 Diopters of myopia. • • • History of intraocular surgery (for example, but not limited to cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months.
* Current or any history of confirmed diagnosis of glaucoma (for example, but not limited to glaucomatous VF changes or nerve changes, or history of glaucoma filtering surgery). e. Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy.
* History or current evidence of ocular disease that, in the opinion of the investigator, may confound assessment of visual function.
* The following medications and treatments are prohibited as they can affect progression of retinal pigmentosa. The participant must not have received or planning to receive the following treatments.
* Any use of ocular stem cell or gene therapy.
* Any treatment with ocriplasmin.
* Treatment with Ozurdex (dexamethasone), Iluvien or Yutiq (fluocinolone 404 acetonide) intravitreal implant.

The following medications and treatments are excluded within the specified timeframe:

* Treatment with an ophthalmic oligonucleotide within the last 9 months (last treatment date is less than 9 months prior to Screening Visit date).
* Treatment with any other product within five times the expected half-life of the product (time from last treatment date to Screening Visit date is at least 4115 times the half-life of the given product).
* Treatment that can alter visual acuity between Screening and Baseline (e.g., periorbital injections.)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population for GYROS will be patients with gyrate atrophy associated with disease-causing variants in the OAT gene.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Structural Outcome: Characterize Change using Quantitative Measures of Progression of the Area of Preserved Retina | Baseline and every year until study completion (4 years)
  Measured by Wide Field Fundus Autofluorescence (FAF)
Structural Outcome: Characterize Change using Quantitative Measures of Progression of the Area of Preserved Retina (Use with FAF for assessments) | Baseline and every year until study completion (4 years)
  Measured by wide field color photography
Metabolic Outcome: Characterize Change in Plasma Ornithine Level | Baseline and every year until study completion (4 years)
  Obtained by fasting plasma amino acids panel and evaluated by a central lab
Metabolic Outcome: Characterize Change in Blood Spot Ornithine Level | Baseline and every 4 months until study completion (4 years)
  Obtained by fasting blood spot test amino acids panel and evaluated by a central lab

SECONDARY OUTCOMES:
Structural Outcome: Ellipsoid zone (EZ) area | Baseline and every year until study completion (4 years)
  Measured by Spectral Domain Optical Coherence Tomography (SD-OCT)
Structural Outcome: Area of Post Subcapsular Cataract | Baseline and every year until study completion (4 years)
  Measured by Red Reflex Photography
Structural Outcome: Foveal Avascular Zone (FAZ) Area and Macular Vessel Density | Baseline and every year until study completion (4 years)
  Measured by OCTA Ancillary Test at Subset of Sites
Functional Outcome: Visual Field Sensitivity Measured with Quantitative Topographic Analysis (Hill of Vision) | Screening visit and every year until study completion (4 years) with the exception of baseline.
  Measured by Octopus 900 Pro
Functional Outcome: Early Treatment of Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score | Screening visit and every year until study completion (4 years) with the exception of baseline.
  Measured on the Electronic Visual Acuity (EVA) system or ETDRS charts.
Functional Outcome: Low Visual Acuity Test - for participants unable to see ETDRS letters | Screening visit and every year until study completion (4 years) with the exception of baseline.
  Measured on the Berkeley Rudimentary Vision Test (BRVT)
Functional Outcome: ETDRS Best Corrected Low Luminance Visual Acuity Letter Score | Screening visit and every year until study completion (4 years) with the exception of baseline.
  Measured on the Electronic Visual Acuity (EVA) system or ETDRS charts.
Functional Outcome: Change in Mean Retinal Sensitivity | Baseline and every year until study completion (4 years)
  Measured by Fundus-Guided Microperimetry (MP)
Functional Outcome: Change in Full-Field Retinal Sensitivity | Baseline and every year until study completion (4 years)
  Measured by full-field stimulus threshold (FST) testing to blue, white, and red stimuli
Functional Outcome: Change in Retinal Function | Baseline and every year until study completion (4 years)
  Measured by full-field electroretinogram (ERG) amplitudes and timing in response to rod- and cone-specific stimuli.
Metabolic Outcome: Proline, lysine, glutamine, glutamate, arginine, and related metabolite: creatine and its precursor guanidinoacetate | Two (2) fasting plasma samples collected on two (2) different days, within ten (10) days of Baseline Visit date and every year until study completion (4 years)
  Obtained by fasting plasma amino acids panel and evaluated by a central lab
Metabolic Outcome: Level of dietary protein control | Baseline and every year until study completion (4 years)
  Obtained from serum albumin sample evaluated by a central lab

OTHER OUTCOMES:
Patient Reported Outcomes Adults 18 years or older | Baseline and every two years until study completion (4 years)
  Measured by Michigan Retinal Degeneration Questionnaire (MRDQ) Visual Symptom and Impact Outcomes Patient Reported Outcome (ViSIO-PRO) Patient-Reported Outcomes Measurement Information System (PROMIS®-29)
Patient Reported Outcomes Adolescents 12-17 years | Baseline and every two years until study completion (4 years)
  Measured by Visual Symptom and Impact Outcomes Patient Reported Outcome (ViSIO-PRO) L. V. Prasad-Functional Vision Questionnaire (LVP-FVQ II)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep S. Singh, MD, Study Chair — John Hopkin's - Wilmer Eye Institute; David Valle, MD, Study Chair — John Hopkin's - Wilmer Eye Institute
Locations (11):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins University, Wilmer Eye Institute, Baltimore, Maryland
  - Harvard Univ., Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania
- INRET Clínica e Centro de Pesquisa, Belo Horizonte, Minas Gerais, Brazil
- University of Toronto, Hospital for Sick Children, Toronto, Ontario, Canada
- Helsinki University Hospital, Helsinki, Finland
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, INSERM-DGOS CIC1423, Paris, France
- University of Tuebingen, Centre for Ophthalmology, Tübingen, Germany
- Vista Vision Eye Clinic, Brescia, Italy
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data will be transmitted to and stored at the FFB Consortium Coordinating Center, under the supervision of Allison Ayala, for use by other researchers including those outside of the study.
Supporting Information: Study Protocol, ICF
Time Frame: After manuscript is published
Access Criteria: Users accessing data must enter an email address

REFERENCES:
- See also: Foundation Fighting Blindness Public Website — https://public.jaeb.org/ffb

DOCUMENTS (2):
  • Study Protocol: Protocol Administrative Change Letter (PACL) (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT05312736/Prot_001.pdf
  • Study Protocol: Gyrate Atrophy Ocular and Systemic Study (GYROS) (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT05312736/Prot_002.pdf